CLINICAL TRIAL: NCT03310593
Title: A Double-blind, Randomized, Placebo-controlled Clinical Trial of Adjunctive Cannabidiol for Bipolar Depression
Brief Title: Cannabidiol as an Adjunctive Treatment for Bipolar Depression
Acronym: CBDBD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: It was interrupted due to the coronavirus pandemic outbreak.
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 63811317300005327
Record Dates: First submitted 2017-06-15; First posted 2017-10-16 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar Affective Disorder
Keywords: bipolar disorder; bipolar depression; cannabidiol; endocannabinoids
MeSH Terms: conditions — Bipolar Disorder | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized and placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Cannabidiol 150-300mg per day for 12 weeks.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Cannabidiol comparator for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol as active intervention.
  Arms: Cannabidiol
Drug: Placebo — Placebo intervention.
  Arms: Placebo

SUMMARY:
Depressive symptoms are associated with significant psychosocial impairment. However, current treatments of bipolar depression are only partially effective.

Cannabidiol is a natural component of cannabis without psychotomimetic or addictive properties. Cannabidiol has been shown to produce therapeutic effects including anticonvulsive, anxiolytic, antipsychotic and neuroprotective effects. The investigators hypothesize that treatment with cannabidiol will result in improvement of depressive and anxiety symptoms, as well as, improvement in functioning and inflammatory biomarkers. During the clinical trial, subjects will receive study medication (cannabidiol 150-300mg/day) or placebo for a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode as part of bipolar I disorder or bipolar II disorder according to Fifth Edition of Diagnostic and Statistical Manual for Mental Disorders (DSM-5) and are able to provide written informed consent.
* Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 12 and MADRS items 1 (Apparent Sadness) and 2 (Reported Sadness) scores ≥ 2 at baseline.
* Young Mania Rating Scale (YMRS) ≤ 11.
* Currently prescribed lithium or valproic acid and derivates (divalproex sodium, sodium valproate) or atypical antipsychotics at therapeutic dosage for at least 04 weeks before the baseline.
* Females must test negative for pregnancy and must be using adequate birth control measures throughout the study.

Exclusion Criteria:

* Another concurrent mental or behavioral disorder that requires psychiatric attention in the past 6 months.
* Young Mania Rating Scale (YMRS) score > 12.
* Current or past drug sensitivity/intolerance to cannabidiol.
* Substance Use Disorder according to DSM-5 within past 6 months, except for nicotine Substance Use Disorder.
* Clinically significant unstable medical illness, neurological disorders or inflammatory/autoimmune diseases.
* Any autoimmune, inflammatory or neurologic disorders that requires treatment with steroidal anti-inflammatory medications or immunotherapy with biologic drugs.
* Actively suicidal or homicidal risk.
* Females who are pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline Montgomery-Asberg Depression Rating Scale (MADRS) scores. | 08 weeks
  * Change from baseline Montgomery-Asberg Depression Rating Scale (MADRS) scores.
  * Scale range: from 0 to 60.
  * Higher values represent more severe symptoms of depression.

SECONDARY OUTCOMES:
Improvement in clinical global impression. | Up to weeks 08 and 12
  * Change from baseline in Clinical Global Impression(CGI-BP) scores.
  * Scale range: from 1 to 7.
  * Higher values represent more severe symptoms of bipolar disorder.
Improvement in anxiety symptoms | Up to weeks 08 and 12
  * Change from baseline in Hamilton Anxiety Rating Scale (HAMA).
  * Scale range: from 0 to 56.
  * Higher values represent more severe symptoms of anxiety.
Improvement in functioning. | Up to weeks 08 and 12
  * Change from baseline Functioning Assessment Short Test (FAST) scores.
  * Scale range: from 0 to 72.
  * Higher values represent more severe functional impairment.
Improvement in biological rhythms. | Up to weeks 08 and 12
  * Improvement in biological rhythms according to Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN).
  * Scale range: from 0 to 88.
  * Higher values represent more severe symptoms of biological rhythms.
Change in BDNF levels in the blood. | Up to weeks 08 and 12
  Change in brain-derived neurotrophic factor (BDNF) levels in the blood.
Change in inflammatory levels in the blood. | Up to weeks 08 and 12
  Change in inflammatory levels in the blood (cytokines, chemokines and C-reactive protein).
Change in endocannabinoid levels in the blood. | Up to weeks 08 and 12
  Change in endocannabinoid levels in the blood (anandamide and 2-arachidonoylglycerol).
Remission of manic symptoms. | Up to weeks 08 and 12
  * Change from baseline in the Young Mania Rating Scale (YMRS) score.
  * Scale range: from 0 to 58.
  * Higher values represent more severe symptoms of mania.
Change in depressive symptoms | Up to weeks 08 and 12
  * Change from baseline in Hamilton Depression Rating Scale (HAMD) score.
  * Scale range: from 0 to 52.
  * Higher values represent more severe symptoms of depression.
Change in psychotic symptoms | Up to weeks 08 and 12
  * Change from baseline in Brief Psychiatric Rating Scale (BPRS) score.
  * Scale range: from 0 to 108.
  * Higher values represent more severe symptoms of psychosis.
Change in depressive symptoms according to MADRS | Up to week 12
  * Higher values represent more severe symptoms of depression.
  * Scale range: from 0 to 60.
Change in depressive symptoms according to PHQ-9 | Up to weeks 08 and 12
  * Change from baseline in Patient Health Questionnaire (PHQ-9) score.
  * Scale range: from 0 to 27.
Change in oxidative stress markers levels in the blood. | Up to weeks 08 and 12
  Change in oxidative stress markers levels in the blood.

OTHER OUTCOMES:
Side effects | Up to weeks 08 and 12
  * Evaluation of side effects according Udvalg for Kliniske Undersogelser (UKU) side effects rating scale.
  * Scale range: from 0 to 144.
  * Higher values represent more severe side effects associated to medications.

CONTACTS AND LOCATIONS:
Overall Officials: Márcia Kauer-Sant'Anna, MD, PhD, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto JV, Crippa JAS, Cereser KM, Vianna-Sulzbach MF, Silveira Junior EM, Santana da Rosa G, Testa da Silva MG, Hizo GH, Simao Medeiros L, Santana de Oliveira CE, Bristot G, Campos AC, Guimaraes FS, Hallak JEC, Zuardi AW, Yatham LN, Kapczinski F, Kauer-Sant'Anna M. Cannabidiol as an Adjunctive Treatment for Acute Bipolar Depression: A Pilot Study: Le cannabidiol comme traitement d'appoint de la depression bipolaire aigue : une etude pilote. Can J Psychiatry. 2024 Apr;69(4):242-251. doi: 10.1177/07067437231209650. Epub 2023 Nov 3. PMID 37920963